CLINICAL TRIAL: NCT06960057
Title: Exploring Virtual Reality as a Clinical Tool for Blood Pressure Reduction and Assessment of White Coat Hypertension/Effect: A Pre- and Post-Intervention Study With ABPM Validation
Brief Title: Virtual Reality as a Tool to Lower Blood Pressure and Anxiety in Clinic Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Lyle W. Baker, Assistant Professor of Medicine, Medical Director of the Hypertension Center, Mayo Clinic Florida, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 25-000347
Record Dates: First submitted 2025-04-21; First posted 2025-05-07 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-05

CONDITIONS: White Coat Hypertension; Hypertension; Blood Pressure; Anxiety; Virtual Reality Exposure Therapy; Ambulatory Blood Pressure Monitoring; Blood Pressure Disorders
Keywords: White Coat Hypertension; White Coat Effect; Hypertension; Ambulatory Blood Pressure Monitoring; Office Blood Pressure; Virtual Reality; VR Headset; Anxiety Reduction; Stress Reduction; Calming Intervention; Virtual Reality in Medicine
MeSH Terms: conditions — White Coat Hypertension; Hypertension; Anxiety Disorders | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Intervention Model Description: This is a single-arm, pre-post interventional study in which all participants receive the same virtual reality (VR) intervention. Each participant undergoes office blood pressure (OBP) measurement and anxiety assessment both before and after a standardized 5-minute VR session. The study evaluates within-subject changes to determine whether VR exposure affects OBP and anxiety levels in adults that will be undergoing ambulatory blood pressure monitoring (ABPM).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Intervention (Experimental): Participants undergoing ambulatory blood pressure monitoring (ABPM) will receive a 5-minute calming virtual reality (VR) session. Blood pressure and anxiety levels will be measured before and after VR exposure to evaluate its effect on office blood pressure and emotional response in a clinical setting.
  Interventions: Behavioral: Virtual Reality Exposure

INTERVENTIONS:
Behavioral: Virtual Reality Exposure — Participants will be exposed to a standardized 5-minute virtual reality (VR) session using a commercially available VR headset. The session features a calming, immersive environment intended to reduce anxiety and lower office blood pressure (OBP) during a clinical visit. The VR experience is delivered after the return of an ambulatory blood pressure monitoring (ABPM) device and before the final BP measurements are obtained. Blood pressure and anxiety scores are assessed immediately before and after VR exposure.

SUMMARY:
This clinical trial aims to evaluate whether a calming virtual reality (VR) experience can reduce office blood pressure (OBP) and anxiety in adults undergoing ambulatory blood pressure monitoring (ABPM) at Mayo Clinic in Florida.

The main questions it aims to answer are:

1. Does a 5-minute calming VR session reduce office blood pressure in patients with suspected white coat hypertension or white coat effect?
2. Does VR exposure reduce self-reported anxiety levels in the clinical setting?
3. Does VR reduce the difference between home (ABPM) and clinic blood pressure readings?

Participants will:

1. Complete two short electronic surveys (before and after VR exposure) on a clinic-provided device.
2. Undergo a 5-minute virtual reality (VR) relaxation session.
3. Have their blood pressure measured before and after the VR session.

Participation will occur during the participant's scheduled ABPM device return visit and will add approximately 30 minutes to the visit.

This is a single-arm, pre-post interventional study where each participant serves as their own control.

DETAILED DESCRIPTION:
This is a prospective, single-arm, pre-post interventional study designed to evaluate the effect of a calming virtual reality (VR) experience on office blood pressure (OBP), home-clinic BP differences, and self-reported anxiety levels in adults undergoing ambulatory blood pressure monitoring (ABPM) at Mayo Clinic in Florida.

White coat hypertension (WCH) and white coat effect (WCE) are conditions where patients exhibit elevated OBP readings in clinical settings that are not representative of their typical blood pressure levels in non-clinical environments. These conditions can lead to misdiagnosis and unnecessary treatment. ABPM is considered the gold standard for differentiating true hypertension from WCH/WCE. Emerging evidence suggests that virtual reality can reduce anxiety and physiological stress responses, making it a promising tool for improving the accuracy of clinic-based blood pressure assessments.

The study will enroll up to 250 participants, with a target accrual of 200 completed cases. Participants are identified through electronic medical records as individuals scheduled for ABPM. Those who meet eligibility criteria and provide informed consent will participate during a single clinic visit coinciding with the return of their ABPM device.

During the study visit, participants will:

1. Complete a short electronic survey (via REDCap on a clinic-provided device) capturing information about their history of hypertension or white coat hypertension/effect, mental health conditions, use of medications for anxiety or mood disorders, anxiety related to doctor visits, recent caffeine intake, and prior VR experience.
2. Complete two standardized anxiety assessments (the Visual Analog Scale [VAS] for anxiety and the State-Trait Anxiety Inventory-6 [STAI-6]) prior to VR exposure.
3. Undergo three resting office blood pressure (OBP) measurements using an automated blood pressure cuff, with results averaged.
4. Participate in a 5-minute immersive VR session featuring a calming, nature-based environment.
5. Undergo three additional resting OBP measurements after VR exposure, with results averaged.
6. Complete repeat VAS and STAI-6 anxiety assessments following the VR session.
7. Complete a brief post-VR survey evaluating comfort, relaxation, side effects, and overall experience.
8. Permit research staff to review their Mayo Clinic electronic medical record for demographic information, relevant medical history, current medications, office blood pressure readings at the ABPM fitting, and ABPM study results.

The study's primary objective is to assess the change in OBP before and after VR exposure. Secondary objectives include evaluating the change in the home-clinic BP difference and measuring changes in anxiety scores. Exploratory analyses will examine predictors of VR responsiveness, including age, sex, baseline anxiety, and history of mental health conditions

This study is minimal risk. The VR headset used is commercially available and not being evaluated as an FDA-regulated device. Adverse effects from VR are expected to be rare and may include mild dizziness or nausea.

This research seeks to generate evidence on whether VR can be used as a simple, non-invasive tool to reduce OBP and anxiety in patients at risk for WCH or WCE and improve the reliability of in-clinic BP measurements. The findings may inform future strategies for integrating VR into routine hypertension care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Undergoing ambulatory blood pressure monitoring (ABPM) at Mayo Clinic Florida for any clinical indication.
* Able and willing to provide informed consent.

Exclusion Criteria:

* History of epilepsy or seizure disorders.
* Significant cognitive impairment (e.g., dementia, Alzheimer's disease).
* Significant visual impairment that prevents visualization of the VR environment.
* History of vestibular disorders (e.g., Meniere's disease, chronic vertigo).
* Unstable cardiovascular conditions (e.g., myocardial infarction within the past year).
* Chronic hypoxemic respiratory failure requiring supplemental oxygen.
* Cervical spine instability or injuries that could impair safe VR use.
* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Change in Office Blood Pressure (OBP) Before and After VR Exposure | Baseline (pre-VR exposure) and immediately post-intervention (post-VR exposure) during the study visit.
  The primary outcome is the within-subject change in office blood pressure (systolic, diastolic, and mean arterial pressure) measured immediately before and after a standardized 5-minute calming VR session among patients with suspected white coat hypertension (WCH) or white coat effect (WCE). Blood pressure is measured in triplicate using an automated device, with the average of the three readings recorded both pre- and post-VR exposure. Effectiveness will be assessed by comparing pre- and post-VR OBP measurements. Diagnosis of WCH or WCE will be confirmed through ambulatory blood pressure monitoring (ABPM).

SECONDARY OUTCOMES:
Change in Home-Clinic Blood Pressure Difference After VR Exposure | Baseline (average daytime BP from ABPM prior to study visit) and next day follow-up study visit during ABPM device return.
  This outcome compares the home-clinic blood pressure difference (defined as the difference between average daytime ambulatory blood pressure monitoring [ABPM] and in-clinic office BP) before and after VR exposure. The goal is to assess whether VR reduces the magnitude of the difference between ABPM readings and in-clinic measurements.
Change in Visual Analog Scale (VAS) for Anxiety Before and After VR Exposure | Baseline (pre-VR exposure) and immediately post-intervention (post-VR exposure) during the study visit.
  The Visual Analog Scale (VAS) for anxiety is a 0-10 scale where participants rate their current anxiety level. A score of 0 indicates no anxiety and a score of 10 indicates the highest possible anxiety. Higher scores reflect worse anxiety symptoms.
Change in State-Trait Anxiety Inventory-6 (STAI-6) Scores Before and After VR Exposure | Baseline (pre-VR exposure) and immediately post-intervention (post-VR exposure) during the study visit.
  The State-Trait Anxiety Inventory-6 (STAI-6) is a validated six-item questionnaire assessing current (state) anxiety. Each item is scored on a 1-4 Likert scale, with a total possible score ranging from 6 to 24. Higher scores indicate greater anxiety. Units on a scale (6-24).
Patient-Reported Acceptability and Satisfaction with the VR Experience | Immediately post-intervention (post-VR exposure) during the study visit.
  Participants will complete a brief post-intervention survey evaluating their experience with the VR session, including comfort, perceived relaxation, and willingness to use VR in future medical visits.
Incidence of Adverse Effects Related to VR Exposure | Immediately post-intervention (post-VR exposure) during the study visit.
  Any participant-reported side effects during or immediately following the VR session (e.g., dizziness, nausea, eye strain, anxiety) will be recorded. Staff will monitor participants throughout the session and document any discomfort or early discontinuation of VR.

CONTACTS AND LOCATIONS:
Overall Officials: Lyle W Baker, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Hypertension. 2018 Jun;71(6):e13-e115. doi: 10.1161/HYP.0000000000000065. Epub 2017 Nov 13. No abstract available. PMID 29133356
- [Background] Pickering TG, Shimbo D, Haas D. Ambulatory blood-pressure monitoring. N Engl J Med. 2006 Jun 1;354(22):2368-74. doi: 10.1056/NEJMra060433. No abstract available. PMID 16738273
- [Background] Freeman D, Reeve S, Robinson A, Ehlers A, Clark D, Spanlang B, Slater M. Virtual reality in the assessment, understanding, and treatment of mental health disorders. Psychol Med. 2017 Oct;47(14):2393-2400. doi: 10.1017/S003329171700040X. Epub 2017 Mar 22. PMID 28325167
- [Background] Ma H, Bian Y, Wang Y, Zhou C, Geng W, Zhang F, Liu J, Yang C. Exploring the effect of virtual reality relaxation environment on white coat hypertension in blood pressure measurement. J Biomed Inform. 2021 Apr;116:103721. doi: 10.1016/j.jbi.2021.103721. Epub 2021 Feb 22. PMID 33631382
- See also: Can A Five-Minute Virtual Reality Headset Intervention Reduce Blood Pressure In Patients With White-Coat Hypertension? — https://digitalcommons.wku.edu/ijesab/vol16/iss3/249/